CLINICAL TRIAL: NCT06828601
Title: Perioperative Lidocaine Infusions for the Management of Pain From Burn Injury: A Pilot Study to Investigate Analgesic and Opioid Sparing Effects
Brief Title: Perioperative Lidocaine Infusions for the Management of Pain From Burn Injury
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ireana Ng, Assistant Professor, Anesthesiology & Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00018912
Record Dates: First submitted 2024-01-22; First posted 2025-02-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Burn Injury; Lidocaine
MeSH Terms: conditions — Agnosia; Burns | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Lidocaine (Active Comparator): Participant receives IV Lidocaine during surgery. Infusion continues for 48 hours. An initial bolus dose of 1.5 mg/kg ideal body weight (IBW) of IV study infusion will be given at the start of surgery, followed by infusion rate of 2.0 mg/kg/hr IBW intraoperatively.This will be reduced to 1.5 mg/kg/hr IBW postoperatively for 48 hours - once the patient has reached recovery.
  Interventions: Drug: IV Lidocaine
- IV Saline (Placebo Comparator): Participant receives IV Saline (placebo) during surgery. Infusion continues for 48 hours. An initial bolus dose of 1.5 mg/kg ideal body weight (IBW) of IV study infusion will be given at the start of surgery, followed by infusion rate of 2.0 mg/kg/hr IBW intraoperatively.This will be reduced to 1.5 mg/kg/hr IBW postoperatively for 48 hours - once the patient has reached recovery.
  Interventions: Drug: IV Saline

INTERVENTIONS:
Drug: IV Lidocaine — Participant receives IV Lidocaine during surgery. Infusion continues for 48 hours. An initial bolus dose of 1.5 mg/kg ideal body weight (IBW) of IV study infusion will be given at the start of surgery, followed by infusion rate of 2.0 mg/kg/hr IBW intraoperatively.This will be reduced to 1.5 mg/kg/hr IBW postoperatively for 48 hours - once the patient has reached recovery.
  Arms: IV Lidocaine
Drug: IV Saline — Participant receives IV Saline (placebo) during surgery. Infusion continues for 48 hours. An initial bolus dose of 1.5 mg/kg ideal body weight (IBW) of IV study infusion will be given at the start of surgery, followed by infusion rate of 2.0 mg/kg/hr IBW intraoperatively.This will be reduced to 1.5 mg/kg/hr IBW postoperatively for 48 hours - once the patient has reached recovery.
  Arms: IV Saline

SUMMARY:
The purpose of this study is to find out if IV lidocaine infusion decreases the need of opioids, improves pain management, and reduces the risks of developing complications from prolonged opioid use in burn injury participants undergoing wound debridement in the operating room.

Participants will:

* be randomized to receive either an IV Lidocaine treatment or an IV Saline Placebo during their surgery. The IV treatment continues for 48 hours after surgery.
* be asked about their pain and how they're feeling at 4 timepoints during the 48 hours.
* be asked about their pain 2 weeks after surgery.

The participant and medical care providers will both be blinded to what IV treatment is being received.

Researchers will compare the 2 groups to see if IV Lidocaine helps decrease the need of opioids, improves pain management, and reduces the risks of developing complications from prolonged opioid use (this includes opioid tolerance, opioid dependence, and opioid induced hyper-sensitivity to pain).

ELIGIBILITY:
Inclusion Criteria:

* Acute burn patients
* 18 years or older
* <20% Total Body Surface Area
* Wound debridement surgery scheduled at Harborview Medical Center

Exclusion Criteria:

* History of polysubstance use
* Chronic opioid use (MED>40mg for more than 6 weeks)
* Cases where the known clinical standard care would be to keep patient intubated postoperatively
* Cases where the known clinical standard care would avoid IV Lidocaine infusion
* Allergy to amide local anesthetics
* Any elevated risk for local anesthetic systemic toxicity as determined by the study team
* Cardiac arrythmias or cardiovascular instability (e.g. shock)
* Severe renal or hepatic impairment
* Pregnancy
* Local anesthesia will be given by another route (e.g. nerve block)
* Prisoners
* Non-English Speaking/reading

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Study for future larger RCT-Recruitment | Through study completion, an average of 6 months
  Recruitment rate (screening and recruitment of 20 patients over 6 months)
Feasibility of Study for future larger RCT-Preliminary Data | Through study completion, an average of 6 months
  Review of preliminary data for calculation of a sample size, minimum number of subjects needed to enroll in a future RCT for adequate power.
Feasibility of Study for future larger RCT-Acceptability of Intervention | Through study completion, an average of 6 months
  Review of randomization and blinding processes, including both patients and clinical provider's experience
Feasibility of Study for future larger RCT-Data collection | Through study completion, an average of 6 months
  The suitability of the methods for data collection, which are In person visits at 24, 48 & 72hr and likely phone/virtual follow-ups at 2 weeks and 3 months
Feasibility of Study for future larger RCT-Reliability of data | Through study completion, an average of 6 months
  The reliability of data collected for analysis of analgesic efficacy includes review of numerical pain scores, total morphine equivalent dose (MED), Quality of Recovery Scores (QoR-15), and Brief Pain Inventory (BPI). Analgesic efficacy is expressed as the NNT, the number of patients who need to receive the active drug for one to achieve at least 50% pain relief compared with placebo over a 4-6h treatment period.
Feasibility of Study for future larger RCT-Outcomes | Through study completion, an average of 6 months
  Review of current Secondary Outcome to determine if appropriate to become Primary Outcomes for future RCT
Feasibility of Study for future larger RCT-Complete Data collection | Through study completion, an average of 6 months
  Determine completion rate of collected data

SECONDARY OUTCOMES:
Length of Hospital Stay | Up to 50 weeks
  This is calculated from the date admitted to the hospital to the date of hospital discharge.
Adverse effects of lidocaine infusion | 48 hours - During the lidocaine infusion
Total MED | MED assessed at 24-, 48-, and 72-hours post-operatively
  MED=Morphine Equivalent Dose. MED are values that represent the potency of an opioid dose relative to morphine. MED equates the many different opioids into a standard value that is based on morphine and its potency.
Pain Scores | Scores assessed at 24-, 48-, and 72-hours post-operatively
  Pain Scores at rest and at movement provided by participant will be a numerical pain score from 0-10, with 0=no pain and 10-worst pain imaginable.
Quality of Recovery Scores | Assessed 24-, 48-, and 72-hours post-operatively
  The Quality of Recovery-15 (QoR-15) is a patient-reported outcome measurement measuring QoR after surgery and anesthesia. The scale is arbitrary and ranges from 0-150 with 4 severity classes; excellent, good, moderate, and poor recovery.
Brief Pain Inventory (Short Form) | Assessed at 2 weeks post-operatively and at 3 months post-operatively
  The Brief Pain Inventory-Short Form (BPI) is a 9-item self-administered questionnaire which rapidly assesses the severity of pain and it's impact on functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Ireana C Ng, MD, Principal Investigator — University of Washington